CLINICAL TRIAL: NCT05295069
Title: Can Postpartum Depression Be Prevented With Care Provided To Primiparas Using Levine's Conservation Model: Single-Blind Randomized Controlled Experimental Study
Brief Title: Can Postpartum Depression Be Prevented With Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gulsen Eryilmaz, Prof. Dr. Gulsen ERYILMAZ, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AtaturkU-GulsenEryilmaz-001
Record Dates: First submitted 2022-03-09; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Sleep Quality, Depression, Postnatal Care, Single-Blind Method, Fatigue, Social Support
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Fatigue

STUDY DESIGN:
Who Masked: Participant
Masking Description: All participants did not know which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): To reduce postpartum depression among the primiparous puerperal women in the intervention group, and a nursing care program was implemented under the guidance of Levine's model. This program was applied with 7 home visits between the 8th and 80th postpartum days. Face-to-face training and training booklets were provided in home visits. As of the fourth home visit, Pilates exercises were performed.
  Interventions: Behavioral: A nursing care program was applied for the intervention group under the guidance of Levine's conservation model.
- The control group (No Intervention): In the control group women received routine postpartum care. No interventions were conducted other than routine postpartum care.

INTERVENTIONS:
Behavioral: A nursing care program was applied for the intervention group under the guidance of Levine's conservation model. — Face-to-face training and training booklets were provided in home visits. As of the fourth home visit, Pilates exercises were performed.
  Arms: The intervention group

SUMMARY:
This study was designed to eliminate postpartum insomnia and fatigue and reduce the risk of postpartum depression through the maintenance of structural, personal, and social integrity with holistic care under the guidance of Levine's conservation model for primiparous puerperal women who experience fatigue and are at risk of developing depression. : A single-blind pretest-posttest randomized controlled study. Women were called to the hospital on the 7th postpartum day and randomly assigned by a computer program to either the intervention group (n=56) or the control group (n=56). Participants did not know which group they were in.

DETAILED DESCRIPTION:
A nursing care program was prepared for the intervention group under the guidance of Levine's conservation model. This program was applied with 7 home visits between the 8th and 80th postpartum days. Face-to-face training and training booklets were provided in home visits. As of the fourth home visit, Pilates exercises were performed. The women in the control group received routine care. Pretest and posttest data were collected with a personal data sheet, visual analogue scale for fatigue, Postpartum Physical Symptom Severity Scale, Postpartum Sleep Quality Scale, Edinburgh Postpartum Depression Scale, and Postpartum Support Scale.

Sleep quality improved for the primiparous puerperal women of the intervention group. They had reduced postpartum fatigue and increased energy; maintained their structural, personal, and social integrity; and had decreased risk of developing postpartum depression with the holistic care provided (all p<0.001). A negative correlation was detected between the support subscale posttest total score from the Postpartum Support Scale and the posttest scores of the Edinburgh Postpartum Depression Scale for the women of the intervention group (r=-0.303; p<0.05)

ELIGIBILITY:
Inclusion Criteria:

* primiparous;
* reading and understanding Turkish;
* normal term delivery;
* no risky situations during pregnancy or delivery;
* high score (≥65 points) from the Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F),
* score of ≥12 points from the Edinburgh Postpartum Depression Scale (EPDS);
* episiotomy;
* hemoglobin value of at least 10.0 mg/dL;
* no current or past history of psychiatric illness.

Exclusion Criteria:

* inability to communicate
* unwillingness to participate in the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale to Evaluate Fatigue Severity Scores | 1- 7th day after giving birth, Time Frame: 2- postpartum 12th week
  The highest score that can be obtained for the fatigue subdimension is 130 and the lowest score is 0. The highest score that can be obtained from the energy subdimension is 50 and the lowest score is 0. Higher scores on items measuring fatigue and lower scores on items measuring energy indicate that the severity of fatigue is high.
Edinburgh Postpartum Depression Scale Scores | 1- 7th day after giving birth, Time Frame: 2- postpartum 12th week
  The highest score that can be obtained from the scale is 30. A score of 12 or more indicates that the individual is at risk of depression.

SECONDARY OUTCOMES:
The Postpartum Support Scale Scores | 1- postpartum 8th day Time Frame: 2- Postpartum 12th week
  The lowest score that can be obtained from the scale is 0 and the highest score is 238. The higher the total score, the greater the need for support and the greater the support that needs to be received.
the Postpartum Sleep Quality Scale Scores | 1- postpartum 8th day Time Frame: 2- Postpartum 12th week
  The lowest and highest possible scores are respectively 0 and 56. Higher scores indicate lower sleep quality.
The Postpartum Physical Symptom Severity Scale Scores | 1- postpartum 8th day Time Frame: 2- Postpartum 12th week
  Total possible scores range between 0 and 54. Higher scores obtained from this scale indicate higher severity of postpartum physical symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- AtaturkU, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available